CLINICAL TRIAL: NCT01425138
Title: Biologic And Non-biologic Systemic Treatments For Moderate To Severe Plaque Psoriasis: A Systematic Review & Meta-Analysis
Brief Title: Systematic Review And Meta-Analysis Of Psoriasis Treatments.
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: University of Connecticut School of Pharmacy and Hartford Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: A3921142
Record Dates: First submitted 2011-08-26; First posted 2011-08-29 (Estimated); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Psoriasis
Keywords: psoriasis; systematic review; meta-analyses
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Psoriasis: Published data on moderate-to-severe plaque psoriasis.

SUMMARY:
This project involved a systematic literature review of published trials of treatments for moderate-to-severe plaque psoriasis. Data was extracted from the publications on various psoriasis endpoints including the Physician Global Assessment (PGA), Dermatology Life Quality Index (DLQI), and Short-Form 36 (SF-36). A traditional meta-analysis and a mixed treatment comparison was conducted on the extracted data.

DETAILED DESCRIPTION:
This project involved a systematic literature review of published trials of treatments for moderate-to-severe plaque psoriasis. Data was extracted from the publications on various psoriasis endpoints including the Physician Global Assessment (PGA), Dermatology Life Quality Index (DLQI), and Short-Form 36 (SF-36). A traditional meta-analysis and a mixed treatment comparison was conducted on the extracted data. We included all published randomized controlled trials of treatments for moderate-to-severe psoriasis that met the study inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Randomized controlled clinical trials of treatments for moderate-to-severe plaque psoriasis.
* Trials had to evaluate at least one of the following: Physician's Global Assessment (PGA), Dermatology Life Quality Index (DLQI) and/or the Short-Form 36 (SF-36).

Exclusion Criteria:

Observational studies

* Trials that did not report the Physician's Global Assessment (PGA),
* Dermatology Life Quality Index (DLQI) or the Short-Form 36 (SF-36).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Moderate-to-severe plaque psoriasis published trials.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2009-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Physician Global Assessment (PGA)
Dermatology Life Quality Index (DLQI)
Short-Form 36 (SF-36)

SECONDARY OUTCOMES:
No secondary outcomes | No secondary outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921142&StudyName=Systematic%20Review%20And%20Meta-Analysis%20Of%20Psoriasis%20Treatments.